CLINICAL TRIAL: NCT04125056
Title: Bioequivalence Test of Hydronidone Capsules in the Hollow Abdominal State of Chinese Healthy Volunteers
Brief Title: Study on Hydronidone Capsule BE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Continent Pharmaceutical Co, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GNI-F351-1801
Record Dates: First submitted 2019-10-09; First posted 2019-10-14 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-02

CONDITIONS: Healthy
MeSH Terms: interventions — Edible Grain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Experimental): Hydronidone capsules (Specification: 30 mg / capsule）
  Interventions: Drug: Hydronidone Capsule(Specification: 30 mg / grain）
- Control group (Placebo Comparator): Hydronidone capsules (Specification: 15 mg / capsule）
  Interventions: Drug: Hydronidone Capsule(Specification: 15 mg / grain）

INTERVENTIONS:
Drug: Hydronidone Capsule(Specification: 30 mg / grain） — Test group
  Arms: test group
Drug: Hydronidone Capsule(Specification: 15 mg / grain） — Control group
  Arms: Control group

SUMMARY:
The purpose of this study was to compare the hydronidone capsules (specification: 30 mg/particle, test preparation) developed by Shanghai Ruixing Gene Technology corporation with Self reference preparation hydronidone capsule (specification: 15 mg/capsule) Differences in the extent and rate of absorption of healthy male subjects in Fasting state in China. Through the main pharmacokinetic parameters and relative bioavailability, whether the two are bioequivalent, and provide a basis for the registration of the test preparation

ELIGIBILITY:
Inclusion Criteria:

1. Gender: Chinese healthy male subjects;
2. Age: 18 to 65 years old, including 18 and 65 years old;
3. Weight should not be less than 50 kg, body mass index (BMI) in the range of 19 to 26 (including the boundary value) ((BMI) = weight (kg) / height 2 (m2));
4. The subject (or his or her partner) has no pregnancy plan during the trial period and 6 months after the end of the trial and voluntarily adopts effective physical contraception and has no sperm donation or egg donation plan;
5. Before the trial, you have a detailed understanding of the nature, significance, possible benefits, possible inconvenience and potential risks, and volunteered to participate in this clinical trial, to communicate well with the researchers, to comply with the requirements of the entire study, and to sign the written Informed consent.

Exclusion Criteria:

1. (Questions) There are any diseases that may affect the safety of the test or the in vivo process of the drug, including but not limited to: liver, kidney, endocrine, cardiovascular, digestive, neurological, mental, respiratory, neoplastic, immune, skin, blood or Researchers of metabolic systems think that it is not suitable for the past medical history or existing medical history of the test [especially those with cardiovascular disease including cardiovascular disease risk, any gastrointestinal diseases affecting drug absorption (such as irritable bowel syndrome symptoms, bowel) History of disease or inflammatory bowel disease), active pathological hemorrhage (such as peptic ulcer), urticaria, epilepsy, asthma, etc. or other diseases that are not suitable for clinical trials;
2. (Questions)allergies: such as those who are allergic to two or more drugs, food; lactose intolerance;
3. (Questions)Any drug that inhibits or induces liver metabolism of the drug within 28 days prior to taking the study drug (common liver enzyme inducer: barbiturate (the most common phenobarbital), carbamazepine, ammonia Mitt, griseofulvin, methamphetamine, phenytoin, glutamine, rifampicin, dexamethasone; common liver enzyme inhibitors: chlorpromazine, cimetidine, ciprofloxacin, metronidazole Oxazole, chloramphenicol, isoniazid, sulfa drug); or any drug (including Chinese herbal medicine) and health care products used within 14 days before the first dose;
4. (Questions) have special requirements for food, can not comply with a unified diet (such as intolerance to standard foods) or have difficulty swallowing;
5. (Questions)Can not tolerate venipuncture and / or have a history of halo, fainting;
6. (Questions)Overdose (over 8 cups a day, 1 cup = 250mL) tea, coffee or caffeinated beverages during the first three months of screening; or take any caffeine and jaundice from the screening to -1 day admission Food or beverage (such as coffee, tea, chocolate, etc.) and other special dieters that affect the absorption, distribution, metabolism, and excretion of drugs;
7. (Questions)Drinking more than 14 standard units per week for the first 3 months of screening (1 standard unit containing 14 g of alcohol, such as 360 mL of beer or 45 mL of 40% alcohol or 150 mL of wine); or no alcohol during the test period Or study any alcohol-containing product within 24 hours prior to the first administration, and the result of the alcohol breath test is greater than 0.0 mg/100 mL;
8. (Questions)Studying blood donation within 3 months prior to the first dose, including component blood or massive bleeding (greater than 450 mL), or planning to donate blood or blood components during the study period or within 3 months after the end of the study;
9. (Questions)Acute disease occurs prior to the pre-study screening phase or prior to study medication;
10. (Questions)Screened to a food or drink containing inducible or inhibited liver metabolic enzymes (such as grapefruit, mango, dragon fruit, grape juice, orange juice and other flavonoids or citrus glycosides) during admission;
11. (Questions)Those who have undergone surgery within 3 months prior to screening, or who plan to undergo surgery during the study period, and those who have received surgery that affect drug absorption, distribution, metabolism, and excretion;
12. (Questions)History of drug abuse, history of drug abuse; positive urine screening;
13. (Questions)The number of cigarettes per day for the first 3 months of screening is greater than 5, or no tobacco products can be stopped during the trial; those who smoked or used any tobacco products during the screening period, and those with positive nicotine tests;
14. Physical examination during screening, vital sign measurement, electrocardiogram examination, laboratory examination (blood routine, urine routine, blood biochemistry, coagulation function), the investigator judged that the abnormality has clinical significance;
15. Hepatitis B surface antigen positive, or hepatitis C antibody positive, or syphilis antibody positive, or HIV antibody positive;
16. Those who have participated in any other clinical trials within 3 months prior to the trial;
17. The investigator believes that there are any circumstances that may affect the subject's informed consent or follow the protocol, or participate in the trial that may affect the outcome of the trial or its own safety.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2019-03-04 (Actual)

PRIMARY OUTCOMES:
Cmax | up to 12 weeks
AUC | up to 12 weeks
Tmax | up to 12 weeks

SECONDARY OUTCOMES:
λz | up to 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China